CLINICAL TRIAL: NCT02560480
Title: Groin Injuries in Finnish Contact Sports: Prospective 2-year Clinical and Magnetic Resonance Imaging Study
Brief Title: Groin Injuries in Finnish Contact Sports
Acronym: Finngroin
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: Orton Orthopaedic Hospital (Other); Mikkeli Central Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 241/2015
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2019-08

CONDITIONS: Groin Injury
Keywords: groin pain, groin injury, magnetic resonance imaging
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- groin injury (group A): magnetic resonance imaging performed in all athletes with acute or subacute groin injury
  Interventions: Device: magnetic resonance imaging
- control (group B): magnetic resonance imaging performed in selected asymptomatic control athletes
  Interventions: Device: magnetic resonance imaging

INTERVENTIONS:
Device: magnetic resonance imaging — to diagonose groin injury exactly in magnetic resonance imaging

SUMMARY:
The prevalence of acute and chronic groin injuries in athletes is between 5 and 10 %. This observational case-control study follows three contact sport teams (soccer, ice-hockey and bandy) for two years to find out the prevalence and reasons for groin pain. Clinical examination, pain scores and pelvic magnetic resonance imaging (MRI) are performed. Hip and groin questionnaire (HAGOS) is used to determine severity of groin injuries.

DETAILED DESCRIPTION:
The prevalence of chronic groin pain in athletes and physically active adults is between 5 and 10 %. Common causes include adductor tendonitis, musculus rectus abdominis tendopathy, osteitis pubis (edema on MRI scans at pubic symphysis) or disruption of the posterior wall of inguinal canal or iliopsoas muscle. This observational case-control study follows three contact sports team (male soccer, ice-hockey and bandy) for two years to find out prevalence of acute and chronic groin pain. Adult (>18 years old) male athletes with acute or chronic groin pain during the study pediod are included. Outcome measures are clinical examination, pain scores, exact diagnosis and repeated pelvic MRI (two times) are performed in each patients and three control atheletes in each team. Hip and groin questionnaire (HAGOS) is used to determine the severity of groin injuries. The end-points of study are prevalence of groin injuries and exact diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* acute (1-30 days) groin injury
* subacute or chronic groin injury (lasting >30 days)
* pain in the groin or hip area

Exclusion Criteria:

* inguinal hernia
* postoperative pain
* metallic plates or screws in the pelvis (MRI impossible)

Ages: 16 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: three contact sport teams (male ice-hockey, soccer, bandy)
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-08; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
prevalence of acute groin injury | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hannu EK Paajanen, MD, Principal Investigator — Department of Surgery, Kuopio Iniversity Hospital, Finland
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

REFERENCES:
- [Derived] Paajanen H, Hermunen H, Ristolainen L, Branci S. Long-standing groin pain in contact sports: a prospective case-control and MRI study. BMJ Open Sport Exerc Med. 2019 Mar 19;5(1):e000507. doi: 10.1136/bmjsem-2018-000507. eCollection 2019. PMID 31191965